CLINICAL TRIAL: NCT04438525
Title: Is the BAT Inhibition Able to Replace Sting Challenges?
Brief Title: Is the BAT Inhibition Able to Replace Sting Challenges? (BATIRS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 30-381 ex 17/18 (BATIRS)
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-11

CONDITIONS: Vespid Venom Allergy
MeSH Terms: interventions — Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- early maintenance phase (Active Comparator): patients who reached the maintenance dose of venom immunotherapy one week (max. +3 weeks) before recruitment will be sting challenged
  Interventions: Diagnostic Test: sting challenge
- maintenance phase (Active Comparator): patients who reached the maintenance dose of venom immunotherapy one year (+/- 2 months) before recruitment will be sting challenged
  Interventions: Diagnostic Test: sting challenge
- after stopping VIT (Active Comparator): patients who finished venom immunotherapy two years (+/- 6 months) before recruitment (duration of VIT: at least 3 years) will be sting challenged
  Interventions: Diagnostic Test: sting challenge
- blood donors (Other): patients with confirmed vespid venom allergy who have not undergone venom immunotherapy (blood donation necessary to perform BAT Inhibition test)
  Interventions: Other: blood donation

INTERVENTIONS:
Diagnostic Test: sting challenge — At the Moment, sting challenges are the only reliable method to identify patients who are not protected by insect venom immunotherapy.
  Arms: after stopping VIT; early maintenance phase; maintenance phase
Other: blood donation — To perform BAT Inhibition Tests, blood samples of patients with confirmed vespid venom allergy, who have not undergone venom immunotherapy, are necessary.
  Arms: blood donors

SUMMARY:
Insect venom allergy is the major cause for severe allergic reactions in Europe. Wasps and honeybees are responsible for the majority of these allergic reactions. Symptoms range from generalized skin symptoms (wheals, swellings) to respiratory or cardiovascular problems such as asthma, dizziness, loss of consciousness, or cardiac arrest. The regular administration of insect venom ('venom immunotherapy') over up to 5 years is a well-established therapy, providing long-term protection from further systemic sting reactions in the majority of patients. However, there is no laboratory test which is able to identify patients who will still react to an insect sting. The only reliable method available is stinging patients with living insects ('sting challenges'). The key issue is that only few centers in Europe perform sting challenges and many patients have no access to these tests. Therefore, it is of utmost importance to find a method which is able to identify patients who are still at risk for future allergic sting reactions.

The inhibition of the basophil activation test (BAT) could be a potential method to monitor the effectiveness of immunotherapy. Basophils are cells which are activated in acute allergic reactions. The basophil activation of blood donors with vespid venom allergy can be measured after adding sera from allergic patients undergoing immunotherapy. In a preliminary study we found that the activation of basophils could be inhibited in all patients treated with vespid venom, however, results must be confirmed in a larger study.

In this study, a total of 219 patients with vespid venom allergy will be included. Those patients who are receiving or who have already finished venom immunotherapy will be sting challenged and blood samples will be taken to perform BAT inhibition experiments. At the same time, donors with confirmed vespid venom allergy, who have not undergone immunotherapy, will be recruited for a blood donation, which is necessary for the BAT inhibition tests.

If results of the preliminary study could be confirmed, the BAT inhibition will facilitate monitoring the effectiveness of venom immunotherapy and patients would benefit from an early detection of lacking tolerance and consequently from the increased venom dose preventing future life threatening systemic sting reactions.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent male and female subjects who are currently treated or who have been treated with vespid venom immunotherapy
* Age ≥18 and ≤70 years
* Written consent of the participant after being informed

Exclusion Criteria:

* Pregnancy
* Autoimmune disease
* Uncontrolled cardiovascular disease
* Uncontrolled asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Outcome sting challenge vs. BAT Inhibition test | 4 hours
  The primary endpoint for the study is the inhibition of the CD63 basophil response (BAT inhibition at a concentration of 11ng/ml) in vespid venom allergic patients. A minimum activation of 25% is required to see sufficient inhibition of basophil activity. Immunotherapy will be considered successful if the BAT inhibition (with added serum) is reduced by at least 80% compared to 'no serum'.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology and Venerology, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No